CLINICAL TRIAL: NCT00422864
Title: A Single-Arm Prospective Trial Evaluating The Local And Systemic Benefits Of Oxaliplatin And 5FU With Concurrent Radiation In Patients With Metastatic Rectal Cancer
Brief Title: A Single Arm Trial of Oxaliplatin and 5FU With Concurrent Radiation in Patients With Metastatic Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sam Ngan, Peter MacCallum Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/35
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: oxaliplatin — Week 1: Oxaliplatin 100 mg/m2 Day 1 (over 2 hours), leucovorin 200mg/m2 Day 1 concurrent with oxaliplatin over 2 hrs (then 5-FU).
  Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day Week 6: as per Week 1, Weeks 8-10: as per Weeks 3-5 Weeks 11: as per Week 1.
Drug: fluorouracil — Week 1: (after Oxaliplatin and leucovorin)5-FU 400mg/m2 bolus Day 1, then 5-FU continuous infusion 2.4 g/m2 over 46 hours from Day 1.
  Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day and continuous infusion 5-FU 200 mg/m2/day on the days of radiotherapy, Week 6: as per Week 1, Weeks 8-10: as per Weeks 3-5 Weeks 11: as per Week 1.
Drug: leucovorin — Week 1: Oxaliplatin 100 mg/m2 Day 1 (over 2 hours), leucovorin 200mg/m2 Day 1 concurrent with oxaliplatin over 2 hrs (then 5-FU) Week 6: as per Week 1, Weeks 11: as per Week 1.
Procedure: External beam radiotherapy — Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day and continuous infusion 5-FU 200 mg/m2/day on the days of radiotherapy, Weeks 8-10: as per Weeks 3-5

SUMMARY:
This trial is a single-arm study for patients presenting with both local and metastatic adenocarcinoma of rectum. The aims of the trial are (1) to determine the tolerability rate, and (2) to determine toxicity rates, pelvic and distant response rates in patients with locally advanced rectal cancer in the presence of distant metastasis who are treated with an interdigitating chemotherapy (oxaliplatin/5-fluorouracil [5FU]) and radiotherapy regimen.

DETAILED DESCRIPTION:
* Week 1: Oxaliplatin 100 mg/m2 Day 1 (over 2 hours), leucovorin 200mg/m2 Day 1 concurrent with oxaliplatin over 2 hrs, then 5-FU 400mg/m2 bolus Day 1, then 5-FU continuous infusion 2.4 g/m2 over 46 hours from Day 1.
* Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day and continuous infusion 5-FU 200 mg/m2/day on the days of radiotherapy,
* Week 6: as per Week 1,
* Weeks 8-10: as per Weeks 3-5
* Weeks 11: as per Week 1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously untreated and pathologically proven adenocarcinoma of the rectum with distant metastasis who would benefit from combined local therapy and systemic chemotherapy.
2. Lower border of tumour must be within 15cm of anal verge.
3. Age >= 18 years.
4. ECOG Performance Status 0-2
5. Absolute Neutrophil Count > 1.5x10^9/L, haemoglobin > 100 g/L, and platelets > 100x10^9/L.
6. Renal: Creatinine clearance >= 55 mL/min (using radioisotope renal scan or derived from serum creatinine using the Cockcroft-Gault formula).
7. Bilirubin <= 2.0 x upper limit of normal.
8. ALT <= 5 x upper limit of normal
9. Life expectancy in excess of 3 months.
10. No symptomatic peripheral neuropathy > grade 2.
11. Males or non-pregnant, non-lactating females. Female patients of child-bearing potential, not surgically sterilized, must use an adequate form of contraception (oral contraceptive pill or barrier method).
12. Signed informed consent

Exclusion Criteria:

1. Prior pelvic radiotherapy
2. Febrile intercurrent illness or infection.
3. History of myocardial infarction within the previous six months or unstable cardiac disease or any other medical condition likely to compromise the safe delivery of chemotherapy or radiotherapy.
4. Concurrent treatment with other anti-cancer therapy.
5. Significant medical conditions which in the opinion of the investigator would compromise the planned delivery of the chemotherapy and radiotherapy or which may be potentially exacerbated by these modalities.
6. Locally recurrent rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Tolerability rate | as per protocol

SECONDARY OUTCOMES:
Toxicity rates | as per protocol
Pelvic response rate | as per protocol
Distant response rate | as per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ngan, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Michael Michael, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCaluum Cancer Centre, Melbourne, Victoria, Australia